CLINICAL TRIAL: NCT06874699
Title: On-campus Supervised Physical Activity Programme for University Students Facing Mental Health Challenges: a Feasibility Study Exploring Feasibility, Acceptability, Fidelity and Preliminary Effects
Brief Title: Evaluation of the Exercise for Wellbeing Pathway at York St John University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York St John University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETH2425-0237
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Mental Health
Keywords: Exercise; Physical activity; Anxiety; Psychological distress; Depression; University student
MeSH Terms: conditions — Psychological Well-Being; Motor Activity; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): This group will comprise of university students who are enrolled on the Exercise for Wellbeing pathway and who have consented to participate in this evaluative study.
  Interventions: Behavioral: Physical activity programme

INTERVENTIONS:
Behavioral: Physical activity programme — The physical activity programme will have the following features:
  * 6-week programme
  * 1-2 supervised physical activity sessions per week
  * 60 minutes per session, including a mixture of physical activities (e.g. walking, other aerobic physical activity, resistance, balance and stretching exercises)
  * Self-selected physical activity intensity
  * Group-based (maximum of 10 students per session)
  * Sessions supervised by a qualified exercise instructor. A member of the University's Wellbeing team will also be present to offer students mental health support, if needed.
  * Physical activity behavioral strategies incorporated into the 6-week programme (e.g., goal setting, action planning, exploring barriers and enablers, setting cues or prompts for self-directed PA)
  * Encouragement to be physically active away from the supervised sessions

SUMMARY:
In autumn 2024, York St John University launched a physical activity programme for university students facing mental health challenges. The purpose of this project is to conduct a mixed-methods evaluative study of this new service over a 6-month period. It is anticipated that 20-40 students will be recruited to the study, which will assess the following: assess the following: feasibility, the extent to which the service can be delivered successfully; acceptability, the extent to which the service is considered appropriate, satisfactory, or attractive by programme recipients and intervention delivery staff; fidelity, the extent to which the key service components (e.g., assessment procedures, physical activity programme) were implemented as planned and adaptations were made; preliminary effects, with relation to physical, mental and social health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Student enrolled at York St John University
* Age 18 years and over
* Undertaking a course which requires attendance at York St John University's Lord Mayor's Walk Campus
* Presenting to the student wellbeing team with mild-to-moderate mental health concerns (defined as experiencing symptoms of poor mental health such as feeling depressed or socially isolated, prolonged stress and anxiety, or experiencing academic decline that makes their daily life more difficult but maintain daily functioning) and expressing an interest in enhancing their mental health and daily functioning

Exclusion Criteria:

* Unwilling or unable to provide written informed consent
* Unable to attend (or to participate in) the scheduled physical activity sessions
* Unsuccessful physical activity clearance using the physical activity readiness questionnaire (PAR-Q+)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | Over the course of the 6-month enrollment period
  The average number of participants recruited per month
Rate of retention | From enrollment to the end of intervention at 6 weeks
  The proportion of participants who complete the study
Rate of attendance | From enrollment to the end of intervention at 6 weeks
  Median number of supervised physical activity sessions attended amongst all participants
Acceptability of the service | At the 6-week follow-up assessment
  The extent to which the service is considered appropriate, satisfactory, or attractive by programme recipients and intervention delivery staff. Assessed primarily via one-to-one interviews and an exit survey.

SECONDARY OUTCOMES:
Fidelity | From enrollment to the end of intervention at 6 weeks
  The extent to which the key service components (e.g., assessment procedures, physical activity programme) were implemented as planned and adaptations were made. Assessed primarily via session record data and post-intervention interviews with participants and service delivery staff.
Mean time per day in moderate-to-vigorous physical activity | Assessed at baseline and at the 6-week follow-up
  Assessed using an Axivity AX6 wrist-worn accelerometer worn continuously for 7 days at each study timepoint
10-item Recovering Quality of Life (ReQoL) questionnaire | Assessed at baseline and at the 6-week follow-up
  The minimum index score for ReQoL-10 is 0 and the maximum is 40, where 0 indicates poorest quality of life and 40 indicates highest quality of life.
9-item Patient Health Questionnaire (PHQ-9) | Assessed at baseline and at the 6-week follow-up
  The total score ranges from 0 to 27 with higher scores indicating more severe depression.
38-item Mental Health Inventory (MHI-38) | Assessed at baseline and at the 6-week follow-up
  All the MHI items are scored on a six-point scale (1-6) except for items 9 and 28, which are scored on a five-point scale (1-5). The raw score range is 38-226, with higher scores on the Mental Health Index indicating less psychological distress and greater psychological well-being.
Resting blood pressure (automated) | Assessed before and after the 6-week intervention period
Estimated maximal oxygen uptake (YMCA submaximal cycle test) | Assessed before and after the 6-week intervention period
Grip strength (Jamar handgrip dynamometer) | Assessed before and after the 6-week intervention period
Lower-limb muscular strength/endurance (30-s sit-to-stand test) | Assessed before and after the 6-week intervention period
Adverse events | From enrollment to the end of the exit assessment after the end of the 6-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Professor Garry Tew, PhD, Principal Investigator — York St John University
Locations (1):
- York St John University, York, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised IPD may be shared on the University's data repository, RaYDaR.

REFERENCES:
- See also: Webpage that describes the University's Exercise for Wellbeing pathway — https://www.yorksj.ac.uk/wellbeing-and-welfare/wellbeing-support/exercise-for-wellbeing/